CLINICAL TRIAL: NCT00465621
Title: Dose Response Study of AL-37807 Ophthalmic Solution in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: C-06-10
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-angle glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

INTERVENTIONS:
Drug: Xalatan

SUMMARY:
The purpose of thie study is to compare the safety and IOP-lowering efficacy of AL-37807 Ophthalmic Solution 0.05%, 0.1% and 0.2% dosed QD AM to Xalatan dosed QD PM and Vehicle in patients with open-angle glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma
* ocular hypertension

Exclusion Criteria:

- VA worse than 0.60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-03; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Mean IP Change from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Study Director — Alcon Research
Locations (1):
- Atlanta, Atlanta, Georgia, United States